CLINICAL TRIAL: NCT05261269
Title: A Dose-escalation Study of the Safety and Pharmacology of DAN-222 in Subjects With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dantari, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DAN-22220205
Record Dates: First submitted 2022-02-15; First posted 2022-03-02 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: HER2-negative Metastatic Breast Cancer
MeSH Terms: interventions — niraparib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (DAN-222) (Experimental): The starting dose of DAN-222 will be administered IV every week (QW) to subjects in the first cohort.
  Interventions: Drug: DAN-222
- Dose Escalation (DAN-222 + niraparib) (Experimental): The starting dose of DAN-222 will be administered IV every week (QW), in combination with daily oral niraparib.
  Interventions: Drug: DAN-222; Drug: Niraparib

INTERVENTIONS:
Drug: DAN-222 — Administered IV every week to subjects
Drug: Niraparib — Administered orally once daily
  Arms: Dose Escalation (DAN-222 + niraparib)

SUMMARY:
This was an open-label, multicenter, dose-escalation study designed to assess the safety, tolerability, and PK of IV administered DAN-222 followed by a dose-escalation of DAN-222 in combination with niraparib:

* Part A is dose escalation of single agent DAN-222
* Part B is dose escalation of DAN-222 in combination with niraparib

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically documented, metastatic, HER2-negative breast cancer that has progressed after two prior lines of therapy (including adjuvant therapy if progressed within the last 12 months, and aromatase inhibitors will be considered a line of therapy). Subjects with HR+ disease can have prior CDK4/6 inhibitors and subjects with BRCAm disease may have prior PARPi therapy. HER2 positivity is defined by standard of care fluorescence in situ hybridization (FISH) and/or 3+ staining by immunohistochemistory (IHC) according to the American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) Clinical Practice Guideline Focused Update.
2. A minimum of 2 weeks or 5 half-lives (whichever is longer) will be required from any prior therapy for mBC, including chemotherapy, immunotherapy and/or radiation therapy.
3. Subjects must have measurable disease as per RECIST v1.1.
4. Females, age 18 years or older.
5. ECOG performance status ≤ 2.
6. Subjects with previously treated brain metastases (surgery, whole or stereotactic brain radiation) are allowed provided the lesions have been stable for at least 4 weeks and the subject is off steroids for at least 7 days prior to first dose of study treatment, and any neurologic symptoms have returned to baseline (without evidence of progression by imaging using the identical imaging modality for each assessment, either MRI or CT scan).
7. Subjects with brain metastases should not require use of enzyme-inducing antiepileptic drugs (eg, carbamazepine, phenytoin, or phenobarbital) within 14 days before first dose of study treatment and during study. Use of newer antiepileptics that do not produce enzyme induction drug-drug interactions is allowed.
8. Subjects must have normal organ and marrow function as defined below:

   * absolute neutrophil count ≥ 1.5 x 109/L without growth factor support in the last 7 days
   * platelets ≥ 100 x 109/L without growth factor support in the last 7 days
   * hemoglobin ≥ 9 g/dL and no blood transfusion within 4 weeks
   * total bilirubin ≤ 1.5 x the upper limit of normal (ULN) (unless Gilbert's Disease)
   * AST(SGOT)/ALT(SGPT) ≤ 2.5 x ULN (≤ 5 x ULN if liver metastases)
   * creatinine clearance ≥ 60 mL/min (calculated using the Cockroft-Gault formula) for subjects with creatinine levels above institutional normal
9. Patients of childbearing potential have a negative serum pregnancy test within 72 hours prior to the first dose of study medication. Non-childbearing potential is defined as (by other than medical reasons):

   * 45 years of age or older and has not had menses for > 1 year
   * Amenorrheic at least 2 years without a hysterectomy and oophorectomy and a follicle stimulating hormone (FSH) value in the postmenopausal range upon pre-study (screening) evaluation
   * Post hysterectomy, bilateral oophorectomy, or tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the subject must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 120 days after the last dose of study therapy.
10. Subject is willing and able to comply with the protocol for the duration of the study including providing medical information, study examinations or tests at scheduled visits and study treatment.

Exclusion Criteria:

1. Any significant medical condition or laboratory abnormalities which place the subject at unacceptable risk if he/she were to participate in the study at clinician's discretion and not otherwise stated below.
2. For the DAN-222 and niraparib combination cohorts, subjects cannot have known sensitivity to FD&C Yellow No. 5 (tartrazine).
3. Allergic reaction to irinotecan, topotecan, or govitecan.
4. Concurrent administration or received cytochrome P450 3A4 (CYP3A4) enzyme inducers or inhibitors within 2 weeks prior to the first day of study treatment.
5. Subjects taking medications know to prolong the QT interval or associated with torsades de pointes, unless the subject can safely discontinue these medications or change to comparable medications that do not significantly prolong the QT interval, at least 5 half-lives or 7 days (whichever is longer) prior to the first dose of DAN-222.
6. History of myelodysplasia, or has a known additional malignancy that progressed or required active treatment within the last 3 years. Exceptions include non-melanoma skin cancer and carcinoma in situ.
7. Carcinomatous meningitis.
8. Subject is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment.
9. Inability to comply with study procedures or unwilling to use adequate birth control.
10. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia that would limit compliance with study requirements.
11. Subject has a heart-rate corrected QT interval (QTc) prolongation > 470 msec at screening.
12. Any serious social, psychosocial, or medical condition or abnormality in clinical laboratory tests that, in the Investigator's judgment, precludes the subject's safe participation in and through a minimum of 4 cycles of treatment, or which could affect compliance with the protocol or interpretation of results.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-10-11 (Actual)

PRIMARY OUTCOMES:
Incidence and nature of Dose Limiting Toxicities (DLTs) | 3 years
Incidence, nature, and severity of adverse events graded according to NCI CTCAE v5.0 | 3 years
Total exposure (area under the curve) from time 0 to the last measurable concentration (AUC0-last) | 3 years
Maximum observed plasma concentration (Cmax) | 3 years
Minimum observed plasma concentration (Cmin through concentration) | 3 years
Terminal half-life (t1/2) | 3 years
Clearance rate | 3 years
Volume of distribution | 3 years

SECONDARY OUTCOMES:
Objective response per RECIST v1.1, defined as the proportion of patients having a best overall response (BOR) of complete response (CR) or partial response (PR), as determined by Investigator review. | 3 years
Progression-free survival per RECIST v1.1, defined as the time from randomization to documented disease progression or death from any cause, whichever occurs earlier as determined by Investigator review. | 3 years
Disease control rate (DCR) per RECIST v1.1, defined as best overall response of complete response (CR), partial response (PR), or stable disease (SD) as determined by Investigator review. | 3 years
Clinical benefit rate (CBR) per RECIST v1.1, defined as the proportion of patients having a BOR of SD ≥ 6 months, PR or CR as determined by Investigator review. | 3 years
Duration of response, defined as the time from first occurrence of a documented objective response until the time of disease progression, as determined by Investigator review with use of RECIST v1.1, or death from any cause during the study. | 3 years

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA - Parkside Cancer Center, Santa Monica, California
  - H Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Michigan, Ann Arbor, Michigan
  - Saint Luke's Cancer Institute, Jackson, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Magee Women's Hospital, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute/Tennessee Oncology, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No